CLINICAL TRIAL: NCT04043429
Title: Restoration vs. Compensation in Neurovisual Rehabilitation of Visual Field Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Professor, Head of Institute, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRT100
Record Dates: First submitted 2014-09-18; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Hemianopia; Brain Injuries, Traumatic
MeSH Terms: conditions — Hemianopsia; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vision Restoration Training (VRT) (Experimental): home-based rehabilitation program which applies intense light stimulation via a PC-monitor to areas of residual vision with a duration of 1 hour daily/six days a week, subjects are asked to respond via button press upon appearance of light stimuli without eye movements
  Interventions: Behavioral: Vision Restoration Training (VRT)
- Vision Exploration Training (VET) (Active Comparator): home-based rehabilitation program to train eye movements upon visual stimuli presented via a PC-monitor with a duration of 1 hour daily/six days a week, subjects are asked to shift their gaze towards targets and respond via button press upon detection of targets
  Interventions: Behavioral: Vision Exploration Training (VET)

INTERVENTIONS:
Behavioral: Vision Restoration Training (VRT)
  Arms: Vision Restoration Training (VRT)
Behavioral: Vision Exploration Training (VET)
  Arms: Vision Exploration Training (VET)

SUMMARY:
Visual field defects (VFD) are a frequent effect of cerebral lesions especially after posterior cerebral artery stroke. The present study was conducted to compare effects of vision restoration training (VRT) and compensation training (Visual Exploration Training, VET) on visual field performance.

ELIGIBILITY:
Inclusion Criteria:

* Visual field defects after brain damage
* lesion age above 6 months
* documented brain lesions due to ischemic stroke, hemorrhage or tumor demonstrated by computer tomography or by magnet resonance imaging

Exclusion Criteria:

* hemispatial neglect
* complete blindness
* severe psychotic diseases
* serious drug abuse
* chronic degenerative diseases (dementia, multiple sclerosis)
* severe motor impairments
* noticeable low intelligence influencing proper comprehension of diagnostic and training instructions
* considerable impaired vision (visual acuity below 0.1 generated by amblyopia, opacity of cornea or lens, maculopathy and other retinal diseases where vision impairment is expected in the next month (e.g. subretinal neovascularisation, retinitis pigmentosa, diabetic retinopathy)
* inability to fixate due to central scotoma, pathological nystagmus or other forms of fixation disabilities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
High Resolution Perimetry - Detectection performance change before vs. after training (%) | 3 months
Humphrey Field Analyzer (Static Perimetry) - Detectection performance change before vs. after training (%) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Inst. f. Medical Psychology, Univ. of Magdeburg, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication
Access Criteria: Contacting the PI

REFERENCES:
- [Result] Sabel BA, Gudlin J. Vision restoration training for glaucoma: a randomized clinical trial. JAMA Ophthalmol. 2014 Apr 1;132(4):381-9. doi: 10.1001/jamaophthalmol.2013.7963. PMID 24504128